CLINICAL TRIAL: NCT07270575
Title: REsorbable SCaffolds With everolimUs-Elution for the Treatment of Infrapopliteal Artery Disease in Patients With Chronic Limb-threatening Ischemia
Acronym: RESCUE
Status: Not yet recruiting | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: RESCUE
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Chronic Limb Threatening Ischemia; Chronic Limb-Threatening Ischemia
Keywords: CLTI; Critical Limb-Threatening Ischemia; Infrapopliteal artery disease; Peripheral artery disease; Esprit BTK Everolimus Eluting Resorbable Scaffold; Drug-eluting resorbable scaffold; Resorbable vascular scaffold; Real-world evidence study; Patients with infrapopliteal disease; Calcified peripheral artery lesions; Infrapopliteal arteries
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult CLTI patients with infrapopliteal calcified lesions: Adult CLTI patients planned to receive the Esprit BTK™ resorbable scaffold following pre-dilatation with angioplasty balloon.
  Interventions: Device: Esprit BTK™ Everolimus Eluting Resorbable Scaffold from Abbott

INTERVENTIONS:
Device: Esprit BTK™ Everolimus Eluting Resorbable Scaffold from Abbott — The Esprit BTK™ is a bioresorbable vascular scaffold designed for arteries below the knee. It provides temporary support to keep the vessel open while releasing everolimus-an antiproliferative drug that helps prevent excessive tissue growth and reduces the risk of restenosis. As the scaffold delivers the medication, it gradually dissolves, potentially lowering long-term risks associated with permanent stents.
  Other Names: Drug-eluting resorbable scaffold

SUMMARY:
RESCUE is a Europe-wide study that will follow 400 people with critical limb-threatening ischemia (CLTI). It aims to see how well Esprit BTK™ Everolimus Eluting Resorbable Scaffolds work in real-life medical settings. The study focuses on people who have heavily calcified arteries in the infrapopliteal areas of the leg.

These drug-eluting resorbable scaffolds release a medication that helps prevent the inner wall of the blood vessel from thickening after injury or surgery. This can reduce the chance of the artery becoming blocked again (a problem called restenosis), while also giving temporary structural support to the vessel. Over time, the scaffold naturally dissolves in the body, which may lower the long-term risks associated with permanent metal stents.

ELIGIBILITY:
Inclusion Criteria:

1. Rutherford classification category ≥4;
2. Treatment of infrapopliteal lesions with the Esprit BTK everolimus eluting resorbable scaffold system following adequate vessel preparation;
3. Calcification of target lesions must be visible on fluoroscopy or CT-angiography;
4. Patients competent and willing to provide informed consent.

Exclusion Criteria:

1. Minors and other vulnerable populations who may not be able to give informed consent freely or for whom participation is not essential to the study (incapacitated and unconscious individuals, persons deprived of liberty, pregnant and breastfeeding women, etc.);
2. Inadequate inflow (>30% stenosis) following optimization;
3. Insufficient direct outflow (less than 1 run-off vessel);
4. Endovascular procedure(s) on the treatment site within 4 weeks before index procedure;
5. Patients planned to receive an above ankle amputation of the target limb;
6. Patients enrolled in ORACLE (ClinicalTrials.gov ID NCT07270562).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CLTI patients treated with the Esprit BTK everolimus-eluting resorbable scaffold following adequate vessel preparation for infrapopliteal artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2032-04 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Number of lesions free from Clinically-Driven Target Lesion Revascularization (CD-TLR) | 12 months
  Defined as freedom from any endovascular re-intervention to the target lesion (± 10 mm) or surgical bypass performed because of restenosis or occlusion of the target lesion.

SECONDARY OUTCOMES:
CD-TLR-free survival per target lesion | Until the end of the follow-up period of 3 years
  Defined as the time between first index procedure and any endovascular re-intervention to the target lesion (± 10 mm) or surgical bypass performed because of restenosis or occlusion of the target lesion.
Clinical response using Rutherford classification categories | 12, 24, and 36 months
  The Rutherford classification is a clinical scale used to categorize the severity of peripheral arterial disease: Category 0 = asymptomatic; Category 1 = mild claudication; Category 2 = moderate claudication; Category 3 = severe claudication; Category 4 = ischemic rest pain; Category 5 = minor tissue loss; Category 6 = severe tissue loss.
Wound status | 12, 24, and 36 months
  Defined as healing status of the dominant ischemic wound of the target limb (complete, partial, unchanged, worsening).
Freedom from major amputation of the target limb | 12 and 24 months
  Defined as absence of any amputation of the target limb (above ankle).
Amputation-free survival | Until the end of the follow-up period of 3 years
  Defined as time between first index procedure and amputation of the target limb, minor (digital, metatarsal), major below the knee or major above the knee (excluding any amputation planned before the index procedure).
Overall survival | Until the end of the follow-up period of 3 years
  Defined as the time between the first index procedure and death of any cause.
Patient-reported health-related quality-of-life | Baseline, Day 0 (day of procedure), 6-, 12-, 24-, 26-months post treatment
  Measured by Vascular Quality of Life Questionnaire - 6 items (VascuQol-6), which is a short patient-reported outcome measure (PROM), used to assess health-related quality of life in people with PAD. It consists of 6 questions, each scored from 1 to 7, with 1 as the worst possible quality of life and 7 as the best possible quality of life. Higher overall scores reflect better quality of life for patients with PAD.
Frequency and severity of procedural complications and other adverse events | Within 30 days after the index procedure
  Grading according to the classification system of the Cardiovascular and Interventional Radiological Society of Europe.
Frequency of major adverse limb events (MALE) and peri-operative death (POD). | 6 months for MALE; Within 30 days after the index procedure for POD
  MALE include above-ankle amputation in the index limb, major re-intervention on the index limb at 6 months and POD includes perioperative (30-day) mortality.
Clinical response using ankle-brachial index (ABI) | 12, 24, and 36 months
  The ankle-brachial index (ABI) is a non-invasive measure calculated as the ratio of systolic blood pressure at the ankle to systolic blood pressure at the arm. ABI categories commonly used to classify peripheral arterial disease are: >1.40 = non-compressible arteries; 1.00-1.40 = normal; 0.91-0.99 = borderline; 0.41-0.90 = mild to moderate peripheral arterial disease; <0.40 = severe peripheral arterial disease.
Clinical response using toe pressure | 12, 24, and 36 months
  The toe pressure test measures distal limb perfusion by recording systolic pressure at the toe. In CLTI patients, toe pressure ≤30 mmHg is commonly used to indicate severe ischemia, while values >30 mmHg suggest better perfusion.
Clinical response using WIfi (wound, ischemia and foot infection) score | 12, 24, and 36 months
  The WIfI classification is a staging system used to assess CLTI based on wound extent, ischemia severity, and foot infection. Each component is graded from 0 (none) to 3 (severe). Lower WIfI scores indicate a lower risk of limb loss and a lesser urgency for revascularization, whereas higher scores indicate greater disease severity, higher amputation risk, and greater potential benefit from revascularization.
Restoration of normal lumen per target lesion | Immediately upon procedure completion
  Defined as residual stenosis ≤30%, immediately after completion of full planned procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Grözinger, Prof. Dr. med., Study Chair — SLK Kliniken Heilbronn GmbH; Marianne Brodmann, Univ.-Prof. Dr. med., Study Chair — Medizinische Universität Graz; Raghu Lakshminarayan, Dr, Study Chair — Hull University Teaching Hospital; Stefan Müller-Hülsbeck, Prof. Dr. med., Study Chair — DIAKO Krankenhaus gGmBH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filippiadis DK, Binkert C, Pellerin O, Hoffmann RT, Krajina A, Pereira PL. Cirse Quality Assurance Document and Standards for Classification of Complications: The Cirse Classification System. Cardiovasc Intervent Radiol. 2017 Aug;40(8):1141-1146. doi: 10.1007/s00270-017-1703-4. Epub 2017 Jun 5. PMID 28584945